CLINICAL TRIAL: NCT06274801
Title: An Open-label Extension Study Evaluating the Long-term Safety and Efficacy of Seralutinib Orally Inhaled for the Treatment of Pulmonary Arterial Hypertension (PAH)
Brief Title: Open-label Extension Study of Seralutinib in Adult Subjects With PAH (PROSERA-EXT)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GB002, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB002-3102; 2023-506334-75 (EudraCT Number)
Record Dates: First submitted 2024-01-19; First posted 2024-02-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: seralutinib; GB002; PROSERA; PROSERA-EXT
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Seralutinib 90 mg (Experimental): Seralutinib inhaled orally twice per day (BID)
  Interventions: Drug: Seralutinib; Device: Gereic Dry Powder Inhaler

INTERVENTIONS:
Drug: Seralutinib — Capsule containing seralutinib
Device: Gereic Dry Powder Inhaler — Generic dry powder inhaler for seralutinib delivery

SUMMARY:
This open-label extension study will evaluate the long-term safety, tolerability and efficacy of orally inhaled seralutinib in subjects who have completed a previous seralutinib study

DETAILED DESCRIPTION:
The treatment period is planned to run until the market approval of seralutinib or until the study is terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have completed a qualifying last visit in a prior seralutinib PAH study on investigational product (IP) and in accordance with the protocol.
2. Evidence of an informed consent document, signed and dated by the subject, indicating that the subject has been informed of all pertinent aspects of the study prior to initiation of any subject-mandated procedures.
3. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
4. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at enrollment visit before first administration of Investigational Product (IP) in this study.
5. WOCBP who are not abstinent and intend to be sexually active with a non-sterilized male partner must be willing to use a highly effective method of contraception from consent through 30 days following the last administration of IP.
6. Male subjects: Non-sterilized male subjects who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom from consent through 90 days after the last dose of IP.

Exclusion Criteria:

1. Severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or seralutinib administration, unless associated with an ongoing AE and discussed with the Sponsor's medical monitor (MM) (or designee).
2. Have any other condition or reason that, in the opinion of the Investigator, would prohibit the subject from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From baseline to end of study (up to 48 months or availability of commercial product)

SECONDARY OUTCOMES:
Changes in distance achieved on the Six-Minute Walk Test (6MWT) | Baseline to Week 12, 24, 36, 48, and 60, and then every 16 weeks thereafter + 4 weeks post dose up to end of study (up to 48 months or availability of commercial product)
  Δ6MWT from Baseline to End of Study
Changes in NT-proBNP | Baseline to Week 12, 24, 36, 48, and 60, and then every 16 weeks thereafter + 4 weeks post dose up to end of study (up to 48 months or availability of commercial product)
  Change in NT-proBNP from Baseline to End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aranda, MD, Study Director — Gossamer Bio Inc.
Locations (115):
- United States (33):
  - Valley Advanced Lung Diseases Institute, Fresno, California
  - Department of Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - UC Davis Health Medical Center, Sacramento, California
  - Stanford Healthcare, Stanford, California
  - University of Florida Health, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Piedmont Physicians Pulmonary & Sleep Medicine of Buckhead, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Northside Hospital - Atlanta, Atlanta, Georgia
  - UI Health Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - INTEGRIS Cardiovascular Physicians, Oklahoma City, Oklahoma
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple Heart and Vascular Institute (Outpatient Clinic), Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - Nexus Research Center, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Outpatient Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
- Argentina (5):
  - Cardiologia Palermo, Buenos Aires
  - Instituto de Cardiologia de Corrientes Juana Francisca Cabral, Corrientes
  - Instuto de Investigacion Clinicas Quilmes, Quilmes
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Hospital Provincial Dr. Jose Maria Cullen, Santa Fe
- Australia (3):
  - Wesley Research Institute, Auchenflower
  - St Vincent's Hospital (Melbourne), Fitzroy
  - Royal Hobart Hospital, Hobart
- University Hospitals of Leuven (Campus Gasthuisberg), Leuven, Belgium
- Brazil (6):
  - Instituto das Pequenas Missionarias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte
  - Complexo de Prevencao, Diagnostico, Terapia e Reabilitacao Respiratoria - Hospital Dia di Pulmao, Blumenau
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto do Coracao do Hospital das Clinicas da Faculdade de medicina da Universidade de Sao Paulo, São Paulo
  - Nucleo de Gestao de Pesquisa/Hospital Sao Paulo - SPDM/UNIFESP, São Paulo
- Canada (4):
  - Peter Lougheed Center, Calgary
  - London Health Sciences Centre - Victoria Hospital, London
  - University of Ottawa Heart Institute, Ottawa
  - University Health Network, Toronto General Hospital, Toronto
- Chile (2):
  - Centro de Investigacion Clinica UC-CICUC, Santiago
  - Enroll SpA, Santiago
- Colombia (2):
  - Fundacion Abood Shaio, Bogotá
  - Fundacion Neumologica Colombiana, Bogotá
- Czechia (2):
  - Institut klinicke a experimentalni mediciny Klinika kardiologie Ambulance plicni hypertenze, Prague
  - Všeobecná fakultní nemocnice v Praze ll. interní klinika kardiologie a angiologie VFN a 1.LF UK Centrum pro plicní hvpertenzi, Prague
- Aarhus Universiteshospital, Aarhus, Denmark
- France (4):
  - CHU Bicetre, Service de Pneumologie et Reanimation Respiratorie, Le Kremlin-Bicêtre
  - Centre Hospitalier REgional Universitaire de Lille Hopital Cardiologique - Institut Coeur Poumon Service de Cardiologie, Lille
  - CHU de Nice - Hopital Pasteur, Nice
  - CHU de Poitiers, Poitiers
- Germany (6):
  - Zentrum fur Pulmonale Hypertonie, Klinik Ill fur lnnere Medizin (Kardiologie, Pneumologie, lnternistische lntensivmedizin), Herzzentrum der Universitat zu Koln, Cologne
  - Universitatsklinikum Giessen und Marburg GmbH Zentrum fur lnnere Medizin, Med. Klinik und Poliklinik II Studienambulanz fur Pulmonale Hypertonie, Giessen
  - Thoraxklinik Heidelberg gGmbH am Universitätsklinikum Heidelberg Zentrum für pulmonale Hypertonie, Heidelberg
  - Klinikum der LMU Medizinische Klinik und Poliklinik V, Munich
  - Krankenhaus Neuwittelsbach, München
  - Klinikum Würzburg Mitte gGmbH Medizinische Klinik mit Schwerpunkt Pneumologie und Beatmungsmedizin, Würzburg
- Greece (4):
  - "Evangelismos" General Hospital of Athens, 1st Department of Clinical Care and Pulmonary Hypertension Clinic, Athens
  - ATTIKON University Hospital, 2nd Critical Care Department, Athens
  - Onassis Cardiac Surgery Center, Non-Invasive Cardiology Department, Kallithea
  - AHEPA University General Hospital of Thessaloniki, 1st Cardiology Clinic, Thessaloniki
- Mater Misericordiae University Hospital, Dublin, Ireland
- Lady Davis Carmel Medical Center, Haifa, Israel
- Italy (4):
  - IRCCS Azienda Ospedaliero Universitaria Di Bologna - Policlinico S. Orsola-Malpighi - UOC Cardiologia, Bologna
  - Azienda Ospedaliera Dei Colli - Ospedale Monaldi, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - A.O.U. Policlinico Umberto I, Roma
- Japan (7):
  - University of Tokyo Hospital, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Kyorin University Hospital, Mitaka
  - Nagoya University Hospital, Nagoya
  - NHO Okayama Medical Center, Okayama
  - Keio University Hospital, Shinjuku-Ku
  - National Cerebral and Cardiovascular Center, Suita
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania
- Mexico (2):
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Unidad de Investigacion Clinica en Medicina, S.C., Monterrey
- Amsterdam UMC, location VU mc, Amsterdam, Netherlands
- Poland (2):
  - Krakowski Szpital Specjalistyczny Im. Sw. Jana Pawla II, Oddzial Kliniczny Chorob Serca i Naczyn z Pododdzialem Intensywnego Nadzoru Kardiologicznego, Krakow
  - Europejskie Centrum Zdrowia Otwock Sp.zo.o. Szpital im. Fryderyka Chopina Oddzial Kardiologiczny, Otwock
- Portugal (2):
  - Unidade Local de Saude de Santa Maria, E.P.E. Hospital Pulido Valente, Lisbon
  - Unidade Local de Saude de Santo Antonio, E.P.E. Hospital de Santo Antonio, Porto
- Romania (2):
  - Institutul De Urgenta Pentru Boli Cardiovasculare Prof. Dr. C. C. Iliescu Cardiology 2, Bucharest
  - "Niculae Stancioiu" Emergency Heart Institute for Cardiovascular Diseases, Cardiology 1 Department, Cluj-Napoca
- Saudi Arabia (2):
  - King Fahad Medical City, Riyadh
  - King Faisal Specialist Hospital and Research Center, Riyadh
- University Clinical Centre of Serbia, Cardiology Clinic, Belgrade, Serbia
- National Heart Centre Singapore, Singapore, Singapore
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (5):
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario de Toledo, Toledo
- United Kingdom (6):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Golden Jubilee National Hospital, Clydebank
  - Hammersmith Hospital, London
  - Royal Free Hospital, Clinical Research Facility, London
  - Freeman Hospital, Newcastle
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No